CLINICAL TRIAL: NCT02361944
Title: Risk of Oxygen During Cardiac Surgery (ROCS) Trial
Brief Title: Risk of Oxygen During Cardiac Surgery Trial
Acronym: ROCS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Frederic T Billings IV, Assistant Professor of Anesthesiology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 131128; R01GM112871 (NIH)
Record Dates: First submitted 2015-01-30; First posted 2015-02-12 (Estimated); Results first posted 2023-08-14 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Cardiac Surgery
Keywords: oxygen; hyperoxia; reactive oxygen species; oxidative stress; oxidative damage; endothelial function; vascular reactivity; mitochondrial function; surgery; anesthesia; kidney injury; renal failure; delirium; myocardial injury; arrythmia
MeSH Terms: conditions — Hyperoxia; Renal Insufficiency; Delirium; Arrhythmias, Cardiac | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normoxia (Experimental): Oxygen administration to maintain a hemoglobin oxygen saturation of 95-97% or arterial PaO2 80-110 mmHg during surgery.
  Interventions: Drug: Oxygen - normoxia
- Hyperoxia (Active Comparator): Fraction of inspired oxygen 1.0 during mechanical ventilation and 0.8 during cardiopulmonary bypass during surgery.
  Interventions: Drug: Oxygen - hyperoxia

INTERVENTIONS:
Drug: Oxygen - normoxia — Titration of FIO2 to maintain normal hemoglobin oxygen saturation (95-97%)
  Other Names: oxygen
  Arms: Normoxia
Drug: Oxygen - hyperoxia — Administration of 1.0 FIO2 during ventilation and 0.8 or above during cardiopulmonary bypass
  Other Names: oxygen
  Arms: Hyperoxia

SUMMARY:
The investigators will recruit and randomize 200 elective cardiac surgery patients to receive physiologic oxygenation (normoxia) or hyper-oxygenation (hyperoxia) during surgery to test the hypothesis that intraoperative physiologic oxygenation decreases the generation of reactive oxygen species, oxidative damage, and postoperative organ injury compared to hyper-oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Open-heart cardiac surgery, defined as surgery on the heart or aorta that requires sternotomy or thoracotomy.

Exclusion Criteria:

* Current acute coronary syndrome (defined as ST elevation myocardial infarction or non-ST elevation myocardial infarction (troponin leak within 72 hours of surgery or consent +/- EKG changes consistent with myocardial ischemia)).
* Home supplemental oxygen use.
* Preoperative supplemental oxygen requirement to maintain arterial O2 sat of 92%.
* Right to left intracardiac shunt including atrial septal defect and ventricular septal defect with Cor Pulmonale.
* Carotid stenosis defined as >50% stenosis.
* Cardiac surgery that requires intraoperative circulatory arrest, such as aortic arch replacement.
* Current use of hemo- or peritoneal dialysis.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2016-04-05 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2021-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic T. Billings, IV, MD, MSc, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Lopez MG, Pandey AK, Hennessy C, Hughes CG, Absi TS, Shah AS, Shotwell MS, Harrison DG, Billings FT 4th; ROCS Trial Investigators. Effects of Oxygen on Perioperative Vascular Function: A Randomized Clinical Trial. J Am Heart Assoc. 2025 Aug 5;14(15):e041778. doi: 10.1161/JAHA.125.041778. Epub 2025 Jul 17. PMID 40673571
- [Derived] Lopez MG, Shotwell MS, Hennessy C, Pretorius M, McIlroy DR, Kimlinger MJ, Mace EH, Absi T, Shah AS, Brown NJ, Billings FT 4th; ROCS trial investigators. Intraoperative Oxygen Treatment, Oxidative Stress, and Organ Injury Following Cardiac Surgery: A Randomized Clinical Trial. JAMA Surg. 2024 Oct 1;159(10):1106-1116. doi: 10.1001/jamasurg.2024.2906. PMID 39110454
- [Derived] Lopez MG, Pretorius M, Shotwell MS, Deegan R, Eagle SS, Bennett JM, Sileshi B, Liang Y, Gelfand BJ, Kingeter AJ, Siegrist KK, Lombard FW, Richburg TM, Fornero DA, Shaw AD, Hernandez A, Billings FT 4th. The Risk of Oxygen during Cardiac Surgery (ROCS) trial: study protocol for a randomized clinical trial. Trials. 2017 Jun 26;18(1):295. doi: 10.1186/s13063-017-2021-5. PMID 28651648

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 213 patients signed consent. 12 participants were withdrawn prior to randomization. 201 were randomized.
Period: Overall Study
Arm/Group | Normoxia | Hyperoxia
Started | 100 | 101
Completed | 100 | 100
Not Completed | 0 | 1
Not completed — surgery cancellation | 0 | 1

BASELINE CHARACTERISTICS:
Population: 101 participant were randomly assigned hyperoxia. 1 of these participant's surgery was cancelled, and this participant was therefore withdrawn from the study. We do not have baseline characteristics for this participant.
Groups:
- Total: Total of all reporting groups
Arm/Group | Normoxia | Hyperoxia | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [58 to 71] | 64 [60 to 72] | 66 [59 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 34 | 60
  Male | 74 | 66 | 140
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 97 | 99 | 196
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 91 | 92 | 183
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 100 | 100 | 200
Serum Creatinine [Median (Inter-Quartile Range); unit: mg/dl] | 1.04 [0.87 to 1.30] | 1.08 [0.84 to 1.36] | 1.06 [0.86 to 1.33]

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Systemic Oxidative Damage
Description: quantified by measuring F2-isoprostanes isofurans following separation from cardiopulmonary bypass or completion of off-pump coronary artery bypass grafting
Time Frame: separation from cardiopulmonary bypass or completion of off-pump coronary artery bypass grafting (approximately 3-5 hours into surgery and intervention)
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
pg/ml | 69 [54 to 89] | 83 [62 to 108]

2. Primary Outcome: Acute Kidney Injury
Description: quantified by change in serum creatinine concentration
Time Frame: baseline to postoperative day 2
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
mg/dl | -0.01 [-0.16 to 0.19] | 0.01 [-0.12 to 0.19]

3. Secondary Outcome: Vascular Reactivity / Endothelial Function (as Measured by Flow Mediated Dilation)
Description: brachial artery flow mediated dilation assessed when patient arrives in ICU after surgery. brachial artery flow mediated dilation is represented as the percent change in brachial artery diameter following 5 minutes of artery occlusion. The entire assessment takes place at ICU admission.
Time Frame: ICU admission (immediately after arrival in ICU from operating room)
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
percentage change | 4.50 [1.22 to 8.12] | 4.71 [1.80 to 9.68]

4. Secondary Outcome: Mitochondrial Function
Description: mitochondrial function in atrial myocardium estimated by quantifying adenylate kinase at the end of surgery and oxygen intervention
Time Frame: up to 2 days following surgery
Population: Analyzed in subjects with tissue available
Measure: Median (Inter-Quartile Range); unit: Absorbance Units (AU)
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 14 | 14
Absorbance Units (AU) | 1884 [1745 to 2236] | 1936 [1591 to 2078]

5. Secondary Outcome: Number of People With Arrhythmia
Description: defined as any atrial fibrillation following surgery until hospital discharge assessed using continuous telemetry, rhythm strips, and electrocardiograms
Time Frame: from surgery to hospital discharge, average of 6 days following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
Participants | 37 | 46

6. Secondary Outcome: Myocardial Injury or Infarction
Description: plasma concentration of creatine kinase, myocardial band
Time Frame: morning of postoperative day 1
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
ng/ml | 27.2 [11.5 to 58.3] | 24.5 [13.4 to 40.8]

7. Secondary Outcome: Number of People With Stroke
Description: Defined as new deficit on neurologic exam and confirmed with radiologic evidence occurring at any point prior to hospital discharge
Time Frame: from surgery to hospital discharge, average of 6 days following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
Participants | 1 | 2

8. Secondary Outcome: Postoperative Cognitive Dysfunction
Description: Median change scores at the Short Blessed Scale (SBT) administered one-year following surgery. The SBT is a validated rating scale, administered by the clinician, measuring the cognitive performance. Sum Total (range 0-28) with 0 indicating no cognitive impairment and 28 indicating severe cognitive impairment.
Time Frame: up to 18 months following surgery
Population: Assessed in participants available for long-term follow-up who were able to complete cognitive assessments
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 57 | 62
score on a scale | 3 [0 to 6] | 2 [0 to 4]

9. Secondary Outcome: Respiratory Failure
Description: reintubation
Time Frame: from surgery to hospital discharge, average of 6 days following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
Participants | 5 | 1

10. Secondary Outcome: Chronic Kidney Disease
Description: eGFR one year following surgery
Time Frame: 12 months following surgery
Population: eGFR assessed in participants available for long-term follow-up
Measure: Median (Inter-Quartile Range); unit: ml/min/1.73 meters squared
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 57 | 69
ml/min/1.73 meters squared | 63.0 [50.8 to 84.8] | 60.4 [44.3 to 84.4]

11. Secondary Outcome: Inflammation
Description: Estimated by quantifying plasma concentration of plasminogen activator inhibitor-1 (PAI-1)
Time Frame: up to 2 days following surgery
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
ng/ml | 31.08 [25.23 to 40.08] | 36.62 [27.54 to 44.93]

12. Secondary Outcome: Hemolysis
Description: plasma free hemoglobin
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
ng/ml | 388,030 [92,628 to 820,820] | 433,274 [74,034 to 982,853]

13. Secondary Outcome: Reactive Oxygen Species Production
Description: TMH electron spin probe
Time Frame: end of surgery, defined as immediately after separation from cardiopulmonary bypass or completion of off-pump coronary artery bypass grafting (approximately 3-5 hours into surgery and intervention)
Measure: Median (Inter-Quartile Range); unit: Absorbance Units (AU)
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
Absorbance Units (AU) | 165,000 [116,000 to 229,500] | 180,100 [145,792 to 258,900]

14. Secondary Outcome: Acute Brain Dysfunction (Delirium)
Description: The number of participants with acute brain dysfunction as assessed by the Confusion Assessment Method for the ICU (CAM-ICU) twice daily while patients are in the ICU or for first 3 postoperative days.
Time Frame: from surgery to hospital discharge, average of 6 days following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
Participants | 16 | 22

15. Secondary Outcome: Oxygenation and Perfusion (Lactate)
Description: arterial lactate measured from arterial blood collected at ICU admission (immediately after arrival in ICU from operating room)
Time Frame: ICU admission (immediately after arrival in ICU from operating room)
Measure: Median (Inter-Quartile Range); unit: mmol/liter
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
mmol/liter | 1.5 [1.2 to 2.3] | 1.8 [1.3 to 2.9]

16. Secondary Outcome: Acute Kidney Injury, According to KDIGO Criteria
Description: KDIGO acute kidney injury is defined as an increase in SCr ≥ 0.3 mg/dL (≥ 26.5 lmol/L) within 48 hours of surgery or 1.5 to 1.9 times baseline within 7 days of surgery
Time Frame: up to 7 days following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
Participants | 21 | 21

17. Secondary Outcome: Acute Kidney Injury Estimated by Urine Concentration of TIMP-2 IGFBP7
Description: Urinary concentration of [TIMP2]*[IGFBP7] 6 hours after ICU admission
Time Frame: baseline to 2 days following surgery
Measure: Median (Inter-Quartile Range); unit: (ng/ml) squared
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
(ng/ml) squared | 0.224 [0.112 to 0.486] | 0.187 [0.075 to 0.423]

18. Secondary Outcome: Acute Kidney Injury Estimated by Urine Concentration of NGAL
Description: Urinary concentration of neutrophil gelatinase-associated lipocalin (NGAL) 6 hours after ICU admission.
Time Frame: baseline to 2 days following surgery
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
ng/ml | 6.9 [3.0 to 17.5] | 4.8 [2.9 to 14.1]

19. Secondary Outcome: Reactive Oxygen Species Production
Description: CAT1H electron spin probe
Time Frame: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: Absorbance Units (AU)
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
Absorbance Units (AU) | 17,300 [8138 to 30,765] | 17,040 [9788 to 45,865]

20. Secondary Outcome: Oxygenation and Perfusion (SpO2)
Description: hemoglobin O2 saturation summarized using SpO2 data continuously measured and recorded every minute during surgery. We calculated the median SpO2 throughout surgery using all the minute to minute values. For example, if a participant had a 5 hour (300 minutes) long surgery, the participant would have 300 SpO2 measurements. We calculated and report the median of those measurements.
Time Frame: during surgery
Measure: Median (Inter-Quartile Range); unit: percent saturation
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
percent saturation | 97 [97 to 98] | 100 [100 to 100]

21. Secondary Outcome: Oxygenation and Perfusion (PaO2)
Description: partial pressure of oxygen in arterial blood measured from blood sampled at end of surgery, defined as following separation from cardiopulmonary bypass or completion of off-pump coronary artery bypass grafting (approximately 3-5 hours into surgery and intervention)
Time Frame: end of surgery, defined as separation from cardiopulmonary bypass or completion of off-pump coronary artery bypass grafting (approximately 3-5 hours into surgery and intervention)
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
mmHg | 99 [96 to 105] | 377 [332 to 426]

22. Secondary Outcome: Oxygenation and Perfusion (Cerebral Oximetry)
Description: brain hemoglobin oxygenation using near-infrared spectroscopy (NIRS). The median percent changes from baseline (baseline measured at beginning of surgery when probes placed on forehead, prior to intervention) throughout surgery was calculated using cerebral oximetry measurements collected every minute throughout surgery. We calculated the difference between baseline and each measurement throughout surgery. For example, if a participant had a 5 hour (300 minutes) long surgery, the participant would have 300 cerebral oximetry measurements. We calculated and report the median of those measurements.
Time Frame: continuously assessed throughout surgery and recorded each minute
Measure: Median (Inter-Quartile Range); unit: percentage change from baseline
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
percentage change from baseline | -7.2 [-14.4 to -0.2] | 6.0 [0.0 to 14.4]

23. Secondary Outcome: Oxygenation and Perfusion (SvO2)
Description: mixed venous O2 saturation, measured from blood sampled from pulmonary artery sampled at end of surgery, defined as following separation from cardiopulmonary bypass or completion of off-pump coronary artery bypass grafting (approximately 3-5 hours into surgery and intervention)
Time Frame: end of surgery, defined as following separation from cardiopulmonary bypass or completion of off-pump coronary artery bypass grafting (approximately 3-5 hours into surgery and intervention)
Measure: Median (Inter-Quartile Range); unit: percent saturation
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
percent saturation | 68 [65 to 73] | 78 [71 to 83]

24. Secondary Outcome: Oxygenation and Perfusion (Cardiac Index)
Description: cardiac output (normalized to body surface area, i.e., cardiac index)
Time Frame: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: liters/min/meter squared
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
liters/min/meter squared | 2.56 [2.14 to 2.88] | 2.48 [1.96 to 3.14]

25. Secondary Outcome: Vascular Reactivity / Endothelial Function (Peripheral Artery Tonometry)
Description: reactive hyperemia index measured at ICU admission (immediately after arrival in ICU from operating room). The reactive hyperemia index is a number generated by an endopat machine performing peripheral artery tonometry. The index ranges from approximately 1-3, where higher values indicate better vascular reactivity and endothelial function.
Time Frame: ICU admission (immediately after arrival in ICU from operating room)
Measure: Median (Inter-Quartile Range); unit: index
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
index | 1.41 [1.14 to 1.78] | 1.23 [0.91 to 1.65]

26. Secondary Outcome: Vascular Reactivity / Endothelial Function (Tension Wire Myography, Endothelial Dependent Vasodilation, EC50)
Description: Effective concentration for 50% dilation acetylcholine dose response, tension wire myography from arterioles dissected from epicardial fat
Time Frame: tissue collected during surgery when heart is exposed approximately 2 hours into intervention
Measure: Mean (95% Confidence Interval); unit: log Molar
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
log Molar | -6.13 [-6.57 to -5.70] | -5.92 [-6.36 to -5.48]

27. Secondary Outcome: Vascular Reactivity / Endothelial Function (Tension Wire Myography, Endothelial Dependent Vasodilation, Emax)
Description: Maximum percentage of arteriole dilation after increasing doses of acetylcholine measured using tension wire myography of arterioles dissected from epicardial fat. The fat sample was collected during surgery when heart is exposed approximately 2 hours into intervention.
Time Frame: tissue collected during surgery when heart is exposed approximately 2 hours into intervention
Measure: Mean (95% Confidence Interval); unit: percent relaxation
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
percent relaxation | 36.2 [25.5 to 46.9] | 39.5 [24.5 to 51.5]

28. Secondary Outcome: Vascular Reactivity / Endothelial Function (Tension Wire Myography, Endothelial Independent Vasodilation, EC50)
Description: Effective concentration for 50% dilation sodium nitroprusside dose response, tension wire myography from arterioles dissected from epicardial fat
Time Frame: tissue collected during surgery when heart is exposed approximately 2 hours into intervention
Measure: Mean (95% Confidence Interval); unit: log Molar
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
log Molar | -6.95 [-7.37 to -6.53] | -5.75 [-6.21 to -5.29]

29. Secondary Outcome: Vascular Reactivity / Endothelial Function (Tension Wire Myography, Endothelial Independent Vasodilation, Emax)
Description: Maximum percentage of arteriole dilation after increasing doses of sodium nitroprusside measured using tension wire myography of arterioles dissected from epicardial fat. The fat sample was collected during surgery when heart is exposed approximately 2 hours into intervention.
Time Frame: tissue collected during surgery when heart is exposed approximately 2 hours into intervention
Measure: Mean (95% Confidence Interval); unit: percent relaxation
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
percent relaxation | 91.5 [83.8 to 99.2] | 92.6 [82.8 to 102.4]

30. Secondary Outcome: Vascular Reactivity / Endothelial Function (Tension Wire Myography, sGC Activation Vasodilation, EC50)
Description: Effective concentration for 50% dilation cinaciguat dose response, tension wire myography from arterioles dissected from epicardial fat
Time Frame: tissue collected during surgery when heart is exposed approximately 2 hours into intervention
Measure: Mean (95% Confidence Interval); unit: log Molar
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
log Molar | -6.89 [-7.48 to -6.30] | -6.66 [-7.20 to -6.12]

31. Secondary Outcome: Vascular Reactivity / Endothelial Function (Tension Wire Myography, sGC Activation Vasodilation, Emax)
Description: Maximum percentage of arteriole dilation after increasing doses of cinaciguat measured using tension wire myography of arterioles dissected from epicardial fat. The fat sample was collected during surgery when heart is exposed approximately 2 hours into intervention.
Time Frame: tissue collected during surgery when heart is exposed approximately 2 hours into intervention
Measure: Mean (95% Confidence Interval); unit: percent relaxation
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
percent relaxation | 97.1 [92.9 to 101.4] | 96.0 [91.9 to 100.2]

32. Secondary Outcome: Vascular Reactivity / Endothelial Function (PAI-1)
Description: Plasminogen activator inhibitor 1
Time Frame: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
ng/ml | 31.2 [25.2 to 40.1] | 36.6 [27.5 to 44.9]

33. Secondary Outcome: Vascular Reactivity / Endothelial Function (E-selectin)
Description: E-selectin
Time Frame: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Normoxia | Hyperoxia
Number analyzed (Participants) | 100 | 100
ng/ml | 16.4 [11.0 to 19.7] | 16.2 [11.3 to 25.0]

ADVERSE EVENTS:
Time Frame: baseline to one year following surgery
Arm/Group | Normoxia | Hyperoxia
All-Cause Mortality (participants affected / at risk) | 2/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 8/100 | 11/100
Other Adverse Events (participants affected / at risk) | 80/100 | 80/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normoxia (N=100) | Hyperoxia (N=100)
Category: Arrythmia, Pacemaker or Cardiac Arrest (Cardiac disorders) | 3 (3) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — refractory postoperative hypoxia requiring ECMO.
right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
anaphylaxis (Immune system disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Re-accumulation of moderate to large pleural effusion requiring reinsertion of chest tube
Seizure (Nervous system disorders) | 2 (2) | 1 (1)
Surgical complications requiring valve replacement revision (Surgical and medical procedures) | 2 (2) | 0 (0)
Severe postoperative hallucinations (Psychiatric disorders) | 1 (1) | 0 (0) — 4-5 days of vivid dreams and visual and auditory hallucinations
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normoxia (N=100) | Hyperoxia (N=100)
Fever (Immune system disorders) | 9 (9) | 6 (6) — Temperature > 38.0 degrees Celsius
Tachycardia (Cardiac disorders) | 5 (5) | 8 (8) — Heart rate > 120 bpm
Hypotension (Vascular disorders) | 29 (29) | 25 (25) — Mean arterial blood pressure < 60 mmHg
Vasoplegia (Vascular disorders) | 34 (34) | 28 (28) — Norepinephrine dose > 5 ug/min
Decreased cardiac output (Cardiac disorders) | 2 (2) | 5 (5) — Cardiac index < 2.0 L/min/m2
Anemia (Blood and lymphatic system disorders) | 49 (49) | 48 (48) — Hematocrit < 30%
Leukocytosis (Blood and lymphatic system disorders) | 37 (37) | 47 (47) — White blood cell count > 15,000
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Platelet count < 50,000

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT02361944/Prot_SAP_000.pdf